CLINICAL TRIAL: NCT03741595
Title: Visual Stimulus Competition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Daniel R. Coates, Assistant Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001197
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Visual Pathway Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Behavioral: Item spacing

INTERVENTIONS:
Behavioral: Item spacing — Spatial proximity of items to one another

SUMMARY:
In this study, we will use behavioral methods to investigate several types of interactions that occur when visual stimuli conflict, such as when objects are presented nearby to each other, or to separate eyes. We will target purely sensory aspects by using simple geometric shapes: letters and lines. Our outcome measure will be performance thresholds.

DETAILED DESCRIPTION:
Participants will be shown visual stimuli on displays and be asked to identify some aspect of the stimuli: their orientation and/or color, the existence of binocular suppression, etc.

In different blocks, stimuli will be manipulated in different ways to characterize basic aspects of visual processing. For example, the contrast, color, and/or spatial layout of stimuli will be varied.

ELIGIBILITY:
Inclusion Criteria:

* Normal Vision
* English language

Exclusion Criteria:

* Less than 20/20 in either eye
* Vision-affecting abnormalities (amblyopia, keratoconus, etc.)
* Ortho-K lenses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Detection probability | 2 hours
  Ability to detect a target stimulus as a function of flanker proximity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, College of Optometry, Houston, Texas, United States